CLINICAL TRIAL: NCT04450888
Title: Effects of Message Framing and Time Discounting on Health Communication for Optimum Cardiovascular Disease and Stroke Prevention(EMT-OCSP): a Pragmatic,Multi-centre, Observer-blinded,12-month Randomised Controlled Study
Brief Title: Effects of Message Framing and Time Discounting on Health Communication for Optimum Cardiovascular Disease and Stroke Prevention
Acronym: EMT-OCSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); China Stroke Databank Center (Other)
Responsible Party: Principal Investigator, Li He, Professor, West China Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 610041
Record Dates: First submitted 2020-06-11; First posted 2020-06-30 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Disease; Stroke; Primary Prevention
MeSH Terms: conditions — Cardiovascular Diseases; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Model A (Other): Total cardiovascular disease (CVD)-free life expectancy gain in one's remaining life.
  Interventions: Other: The strategic use of messages in risk communication
- Model B (Other): Average CVD-free life expectancy gain per year.
  Interventions: Other: The strategic use of messages in risk communication
- Model C (Other): Total CVD-free life expectancy loss that can be reclaimed in one's remaining life.
  Interventions: Other: The strategic use of messages in risk communication
- Model D (Other): Average CVD-free life expectancy loss that can be reclaimed per year.
  Interventions: Other: The strategic use of messages in risk communication

INTERVENTIONS:
Other: The strategic use of messages in risk communication — The interventions in the EMT-OCSP study are strategic health messages delivered (gain-framed vs.loss-framed and long-term vs.short-term contexts) to individuals based on their calculated CVD-free life expectancy and potential interventional benefits.

SUMMARY:
Effects of Message framing and Time discounting on heath communication for Optimum Cardiovascular disease and Stroke Prevention（EMT-OCSP）is a pragmatic, 2 × 2 factorial, randomized, controlled, observer blinded, multicenter trial with four parallel groups. It aims to determine if risk and intervention communication strategy（gain-framed versus loss-frame, long-term context versus short-term context and the potential interaction）have different effect on optimizing adherence to clinical preventive management （in the endpoint of CVD risk reduction）for subjects with at least one moldable risk factor for CVD.

DETAILED DESCRIPTION:
Scientific title Effects of Message framing and Time discounting on health communication for Optimum Cardiovascular disease and Stroke Prevention(EMT-OCSP): a pragmatic randomised controlled study

Principal Investigator Li He

Study period 2020-07-01-2022-01-21

Hypotheses and aims When communicating cardiovascular disease（CVD）risk to individuals, different presentation of information carries its own connotations and biases. The one or the other pattern of the presentation may affect individuals' decision making.This study aims to determine if risk and intervention communication strategy（gain-framed versus loss-frame, long-term context versus short-term context and the potential interaction）have different effect on optimizing adherence to clinical preventive management （in the endpoint of CVD risk reduction）for subjects with at least one moldable risk factor for CVD. We aim to provide evidence for practitioners regarding messaging strategies that improve communication effectiveness and further reduce the risk of CVD events in the population, as well as to develop more effective communication strategies for groups of people with different characteristics to maximise patient adherence to lifestyle modifications and medical treatment.

Primary outcome Ten-year CVD risk, lifetime CVD risk and CVD-free life expectancy after 1 year according to the LIFE-CVD model.

Secondary outcomes CVD risk factors [blood pressure(BP) and serum cholesterol, low-density lipoprotein (LDL), non-high-density lipoprotein (HDL), triglycerides and fasting glucose levels],lifestyle factors (physical activity, tobacco use, alcohol use and eating habits), pharmacological treatments for hypertension, dyslipidaemia and diabetes, and anti-thrombotic drug prescriptions after 1 year.

Study design The EMT-OCSP trial is designed as a pragmatic, 2 × 2 factorial, randomized, controlled, observer blinded, multicenter trial with four parallel groups. Randomization will be performed as block randomization with a 1:1:1:1 allocation.

Study population and sample size Subjects with at least one moldable risk factor for CVD. The sample size calculations revealed that the enrolment of 15,000 participants would be sufficient, allowing for a 20% drop-out rate.

Follow-up period One year

ELIGIBILITY:
Inclusion Criteria:

* aged 45-80 years,
* personally own and use a smartphone (Apple or Android platform) with Internet access,
* and have at least one of the following CVD risk factors: history of CVD at age < 60 years in a first-degree relative, smoking, diabetes, hypertension, and low-density lipoprotein (LDL)cholesterol ≥ 4.5 mmol/L.

Exclusion Criteria:

* participants with histories of CVD, heart failure, or chronic kidney disease (estimated glomerular filtration rate < 30 mL/min/1.73m2);
* those with terminal malignancy at baseline;
* those with severe psychological or mental disorders
* violation of the study protocol and participation in another clinical study during follow-up

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13114 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
10-year CVD risk | At the 1-year follow-up
Lifetime CVD risk | At the 1-year follow-up
CVD-free life expectancy | At the 1-year follow-up

SECONDARY OUTCOMES:
Changes in systolic and diastolic blood pressure | At the 1-year follow-up
Changes in serum cholesterol level | At the 1-year follow-up
Changes in serum LDL level | At the 1-year follow-up
Changes in serum non-HDL level | At the 1-year follow-up
Changes in serum triglycerides level | At the 1-year follow-up
Changes in fasting glucose level | At the 1-year follow-up
Changes in physical activity (International Physical Activity Questionnaire or International Physical Activity Questionnaire Short Version Modified for Elderly) | At the 1-year follow-up
Changes in tobacco use | At the 1-year follow-up
  Tobacco use status (current, former, never) in the records at visits
Changes in alcohol use (AUDIT questionnaire) | At the 1-year follow-up
Changes in dietary habits (food frequency questionnaire) | At the 1-year follow-up
Changes adherence to pharmacological treatments for hypertension (proportion of persistent medication user） | At the 1-year follow-up
  A persistent medication user is defined as a participant who has purchased the drug at least once during each 3-month interval during our study.
Changes adherence to pharmacological treatments for dyslipidaemia (proportion of persistent medication user） | At the 1-year follow-up
Changes adherence to pharmacological treatments for diabetes (proportion of persistent medication user） | At the 1-year follow-up
Changes adherence to anti-thrombotic therapy (proportion of persistent medication user） | At the 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Li He, M.D., Principal Investigator — West China Hospital
Locations (1):
- Health center of Sipo town, Yibin, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers affiliated with the EMT-OCSP study will have access to an internal webpage listing available aggregated datasets and variables; they will not have access to individual data or the original database.External researchers collaborating with at least one steering group member may submit standardised applications for data via this webpage.Upon steering group approval, the data manager will export anonymised aggregated data to authorised researchers.
Time Frame: 6 months after publication

REFERENCES:
- [Derived] Zhou M, Guo J, Chen N, Ma M, Dong S, Li Y, Fang J, Zhang Y, Zhang Y, Bao J, Hong Y, Lu Y, Qin M, Yin L, Yang X, He Q, Ding X, Chen L, Wang Z, Mi S, Chen S, Zhu C, Zhou D, He L. Effects of Message Framing and Time Discounting on Health Communication for Optimum Cardiovascular Disease and Stroke Prevention (EMT-OCSP): a protocol for a pragmatic, multicentre, observer-blinded, 12-month randomised controlled study. BMJ Open. 2021 Mar 24;11(3):e043450. doi: 10.1136/bmjopen-2020-043450. PMID 33762233